CLINICAL TRIAL: NCT04979364
Title: Transcultural Validation of a French Version of the Prescription Opioid Misuse Idex Scale (POMI-5F)
Brief Title: French Version of POMI Scale
Acronym: POMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: POMI
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain; Opioid Misuse
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
French translation and validation of the Prescription Opioid Misuse Index scale (POMI), a brief questionnaire to assess opioid prescription misuse. In view of the increase in the prescription of opioid analgesics for chronic non-cancer pain (CNCP), this tool is particularly interesting to use during medical consultations to screen misuse in opioids user patients. We conducted an observational, prospective and multicenter psychometric study with a cross-cultural validation in 154 CNCP patients treated by opioid at least from 3 months, in two pain clinics.

DETAILED DESCRIPTION:
Chronic pain prevalence in the general population was estimated at 31% in the world, which makes it a major public health problem, not only because of its enormous impact on patients' quality of life, but also because of its significant economic impact on society, with direct and indirect costs. Despite the lack of scientific evidence demonstrating their long-term benefits, analgesic opioids are largely used for treating chronic non-cancer pain (CNCP) lead to an increase of opioid use in recent decades in developed countries. Indeed, worldwide, opioid analgesic prescription use more than doubled from 2001 to 2013, most signiﬁcantly in North America and in Western and Central Europe. Between years 2004 and 2017 in France, while overall analgesic opioid prescription use in the general population decreased by 8.9%, the used strong opioids increased by 104%. The same finding about increase in the use strong opioids was made in USA, Canada and UK. However, the use of opioid analgesics is not without risk, several international studies showed an increase opioid use disorders, hospitalizations and deaths related to the use of opioid analgesics. In France, rates of prescribed opioid-related hospital admissions increased by 167% from 2000 to 2017 and opioid-related deaths signiﬁcantly increased by 146% (1,3 à 3,2 deaths / 1,000,000 habitants from 2000 to 2015). A similar observation can be made in the United States, where deaths from prescription opioid overdose have risen sharply in recent years, but in a much higher proportion than in France (in 2016 in the U.S., more than 42,000 overdose deaths, or an annual prevalence of 133 deaths/1,000,000 population).

In the context of CNCP, opioid analgesics are subject to increasing misuse in relation to a greater number of prescriptions but also through other sources of obtaining (doctor shopping) hat may contribute to the increase in risks associated with the use of opioid analgesics (hospitalization, death). Few studies in France, assessed the misuse of analgesic opioids, based on the evaluation of "doctor shopping" from healthcare databases, and particularly, Chenaf et al., showed an increase of analgesic opioids shopping behavior by 34%, between 2004 to 0.67% in 2017. It is therefore important to be able to identify analgesic opioid misuse. Actually Prescription Opioid Misuse Index (POMI) scale was validated in 2008 by American team in 137 patients recruited from community substance abuse treatment programs, regional jails, pain clinics and private internal medicine practices.

The primary objective was the cross-cultural validation of French version of an opioid analgesic misuse screening scale (POMI) in chronic pain patients in primary care. The secondary objective was the assessment of the relationship between pain intensity and analgesic opioid misuse.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or more, suffered from chronic non-cancer pain for at least 6 months, with at least one analgesic opioid daily for 3 months, and follow in pain clinic.

Exclusion Criteria:

* inability to read or understand questionnaires alone, cancer, and impossibility to do test and retest questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chonic non-cancer pain.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
psychometric properties of POMI scale | Once. Day 1
  Construct validity, internal consistency, test-retest reliability, and convergent validity of POMI scale French version (POMI-5F).
  POMI scale is a self-evaluation scale with 8 items scored 0 (absence) or 1 (presence). The questionnaire is presented in 8 questions, of which 6 are used to calculate a score which is the sum of positive answers; when this score reaches 2, it's considered as positive and describe a misuse.
psychometric properties of POMI scale | Once. At 2 to 4 weeks (Re-TEST phase)
  Construct validity, internal consistency, test-retest reliability, and convergent validity of POMI scale French version (POMI-5F).
  POMI scale is a self-evaluation scale with 8 items scored 0 (absence) or 1 (presence). The questionnaire is presented in 8 questions, of which 6 are used to calculate a score which is the sum of positive answers; when this score reaches 2, it's considered as positive and describe a misuse.